CLINICAL TRIAL: NCT05276986
Title: Effects of Delayed Muscle Pain on Respiratory Muscle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 10.01.2022
Record Dates: First submitted 2022-01-12; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-01

CONDITIONS: Muscle Soreness; Exercise; Respiratory Muscles; Respiratory Function Tests
Keywords: Muscle Soreness; Exercise; Respiratory Muscles; Respiratory Function Tests
MeSH Terms: conditions — Myalgia; Motor Activity

STUDY DESIGN:
Intervention Model Description: 24 healthy university students (n=11 female, n=13 male) with a mean age of 21±2 years included the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DOMS protocol group (Experimental): DOMS was induced for the trunk muscles with a load equals to 80% of the maximum repetitive voluntary contraction. Pulmonary function parameters, respiratory muscle strength and endurance, exercise capacity, pain, fatigue, and dyspnea perception severity were recorded before DOMS and at the 24th and 48th hours after DOMS.
  Interventions: Other: DOMS protocol

INTERVENTIONS:
Other: DOMS protocol — For a maximum repetition of the trunk muscles, two measurements were made with a 45-second rest interval.The values were recorded in Newtons by taking the maximum value of the two repetitions measured. DOMS was formed by eccentric contraction with 80% of this determined value.To generate DOMS in the trunk, participants were seated on the bench with the knees flexed at 90° and the soles of the feet in full contact with the floor, keeping the weight at 80% of the predetermined maximum repetition.The participants were asked to perform trunk extension with eccentric contraction of the trunk in 5 seconds, and trunk flexion with concentric contraction in 3 seconds.Two-minute rests between sets and 45-second rests between repetitions were given.The date and time of the created DOMS were recorded and the measurements were repeated at the 24th and 48th hours.

SUMMARY:
The aim of the study was to determine whether delayed-onset muscle soreness (DOMS) in trunk muscles has an effect on respiratory function parameters, respiratory muscle strength, respiratory muscle endurance, and exercise capacity.

DETAILED DESCRIPTION:
In 24 healthy university students was induced for the trunk muscles with a load equals to 80% of the maximum repetitive voluntary contraction. Pulmonary function parameters, respiratory muscle strength and endurance, exercise capacity, pain, fatigue, and dyspnea perception severity were recorded before DOMS and at the 24th and 48th hours after DOMS.

After DOMS, there is a decrease in respiratory performance values and exercise capacity of healthy individuals and athletes. Therefore, it should be taken into account that delayed muscle soreness before the competition may affect performance. It may be beneficial to take precautions for delayed muscle pain while creating training and exercise programs, and to create treatment programs in case of the emergence of DOMS.

ELIGIBILITY:
Inclusion Criteria:

* Being a healthy individual between the ages of 18-25
* Not having a regular exercise habit
* No infection until at least 3 weeks before the study

Exclusion Criteria:

* Lung disease
* Cardiovascular disease
* Neurological disease
* Orthopedic disease

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-17 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Tests (FVC) | Pulmonary function test measurements were made in all individuals at baseline.
  Forced vital capacity (FVC) was evaluated. The volume of air that is exhaled quickly and strongly following a deep inspiration. Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used.
Pulmonary Function Tests (FEV1) | Pulmonary function test measurements were made in all individuals at baseline.
  Forced expiratory volume in the first second (FEV1) was evaluated. It is the volume of air expelled in the first second from the start of the forced vital capacity maneuver. It gives information about the restriction on major airlines in general.Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used. Individuals were asked to make a forced expiration after maximum inspiration.
Pulmonary Function Tests (FEF25%-75%) | Pulmonary function test measurements were made in all individuals at baseline.
  Flow rate value of forced expiratory volume (FEF25%-75%) was evaluated. It is the mean flow rate in 50% of the forced vital capacity maneuver. Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used. Individuals were asked to make a forced expiration after maximum inspiration.
Pulmonary Function Tests (VC) | Pulmonary function test measurements were made in all individuals at baseline.
  Vital capacity (VC) was evaluated. It is the volume of air in the lungs that varies between full inspiration and maximum expiration. It is possible to measure the volume of both a slow and vigorous exhalation after a deep inspiration.Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used.
Pulmonary Function Tests (FVC) | Pulmonary function test measurements were made in all individuals at the 24th hours after the trunk-oriented DOMS.
  Forced vital capacity (FVC) was evaluated. The volume of air that is exhaled quickly and strongly following a deep inspiration. Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used.
Pulmonary Function Tests (FEV1) | Pulmonary function test measurements were made in all individuals at the 24th hours after the trunk-oriented DOMS.
  Forced expiratory volume in the first second (FEV1) was evaluated. It is the volume of air expelled in the first second from the start of the forced vital capacity maneuver. It gives information about the restriction on major airlines in general.Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used. Individuals were asked to make a forced expiration after maximum inspiration.
Pulmonary Function Tests (FEF25%-75%) | Pulmonary function test measurements were made in all individuals at the 24th hours after the trunk-oriented DOMS.
  Flow rate value of forced expiratory volume (FEF25%-75%) was evaluated. It is the mean flow rate in 50% of the forced vital capacity maneuver. Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used. Individuals were asked to make a forced expiration after maximum inspiration.
Pulmonary Function Tests (VC) | Pulmonary function test measurements were made in all individuals at the 24th hours after the trunk-oriented DOMS.
  Vital capacity (VC) was evaluated. It is the volume of air in the lungs that varies between full inspiration and maximum expiration. It is possible to measure the volume of both a slow and vigorous exhalation after a deep inspiration.Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used.
Pulmonary Function Tests (FVC) | Pulmonary function test measurements were made in all individuals at the 48th hours after the trunk-oriented DOMS.
  Forced vital capacity (FVC) was evaluated. The volume of air that is exhaled quickly and strongly following a deep inspiration. Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used.
Pulmonary Function Tests (FEV1) | Pulmonary function test measurements were made in all individuals at the 48th hours after the trunk-oriented DOMS.
  Forced expiratory volume in the first second (FEV1) was evaluated. It is the volume of air expelled in the first second from the start of the forced vital capacity maneuver. It gives information about the restriction on major airlines in general.Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used. Individuals were asked to make a forced expiration after maximum inspiration.
Pulmonary Function Tests (FEF25%-75%) | Pulmonary function test measurements were made in all individuals at the 48th hours after the trunk-oriented DOMS.
  Flow rate value of forced expiratory volume (FEF25%-75%) was evaluated. It is the mean flow rate in 50% of the forced vital capacity maneuver. Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used. Individuals were asked to make a forced expiration after maximum inspiration.
Pulmonary Function Tests (VC) | Pulmonary function test measurements were made in all individuals at the 48th hours after the trunk-oriented DOMS.
  Vital capacity (VC) was evaluated. It is the volume of air in the lungs that varies between full inspiration and maximum expiration. It is possible to measure the volume of both a slow and vigorous exhalation after a deep inspiration.Test were performed using a portable spirometer (MIR Spirolab III srl, Italy). During the test, the subject was in a sitting position and their nose was clamped. The test were repeated three times and the best measurement value was used.
Respiratory Muscle Strength Measurement | This test was carried out at baseline.
  Respiratory muscle strength validity and reliability were demonstrated by measuring maximal inspiratory (MIP) and maximal expiratory (MEP) pressures with a portable intraoral pressure measuring device (MicroRPM Respiratory Muscle Testing, Germany). Measurements were made using a clamp that prevents nasal breathing and were performed 5 times until a difference of 5 cmH2O remained, with a 30-second rest period between measurements to record the best value, and the best result was recorded in cmH2O. The recorded values were calculated and recorded with the expected values according to age and gender.
Respiratory Muscle Strength Measurement | This test was carried out at the 24th after DOMS.
  Respiratory muscle strength validity and reliability were demonstrated by measuring maximal inspiratory (MIP) and maximal expiratory (MEP) pressures with a portable intraoral pressure measuring device (MicroRPM Respiratory Muscle Testing, Germany). Measurements were made using a clamp that prevents nasal breathing and were performed 5 times until a difference of 5 cmH2O remained, with a 30-second rest period between measurements to record the best value, and the best result was recorded in cmH2O. The recorded values were calculated and recorded with the expected values according to age and gender.
Respiratory Muscle Strength Measurement | This test was carried out at 48th hours after DOMS.
  Respiratory muscle strength validity and reliability were demonstrated by measuring maximal inspiratory (MIP) and maximal expiratory (MEP) pressures with a portable intraoral pressure measuring device (MicroRPM Respiratory Muscle Testing, Germany). Measurements were made using a clamp that prevents nasal breathing and were performed 5 times until a difference of 5 cmH2O remained, with a 30-second rest period between measurements to record the best value, and the best result was recorded in cmH2O. The recorded values were calculated and recorded with the expected values according to age and gender.
Respiratory Muscle Endurance Test | This test was performed at baseline.
  Respiratory muscle endurance was evaluated with a threshold-loaded (constant) respiratory muscle trainer (Power Breathe®, POWERbreathe International Ltd. Warwickshire, England) with proven validity and reliability . In the evaluation, measurements were made in the upright sitting position in the chair while the nose of the individuals was closed with a clip.
  Initial workload was applied at 60% of the maximal inspiratory pressure. Participants were asked to continue inspiring despite constant inspiratory workload.
  The respiratory muscle endurance value was obtained by multiplying the maximum workload of the test that can be sustained for at least one minute.
  Individuals were told that the test could be terminated if severe fatigue and extreme shortness of breath were experienced during the test.
  The results of the test were recorded.
Respiratory Muscle Endurance Test | This test was performed at 24 hours after DOMS.
  Respiratory muscle endurance was evaluated with a threshold-loaded (constant) respiratory muscle trainer (Power Breathe®, POWERbreathe International Ltd. Warwickshire, England) with proven validity and reliability . In the evaluation, measurements were made in the upright sitting position in the chair while the nose of the individuals was closed with a clip.
  Initial workload was applied at 60% of the maximal inspiratory pressure. Participants were asked to continue inspiring despite constant inspiratory workload.
  The respiratory muscle endurance value was obtained by multiplying the maximum workload of the test that can be sustained for at least one minute.
  Individuals were told that the test could be terminated if severe fatigue and extreme shortness of breath were experienced during the test.
  The results of the test were recorded.
Respiratory Muscle Endurance Test | This test was performed at 48 hours after DOMS.
  Respiratory muscle endurance was evaluated with a threshold-loaded (constant) respiratory muscle trainer (Power Breathe®, POWERbreathe International Ltd. Warwickshire, England) with proven validity and reliability . In the evaluation, measurements were made in the upright sitting position in the chair while the nose of the individuals was closed with a clip.
  Initial workload was applied at 60% of the maximal inspiratory pressure. Participants were asked to continue inspiring despite constant inspiratory workload.
  The respiratory muscle endurance value was obtained by multiplying the maximum workload of the test that can be sustained for at least one minute.
  Individuals were told that the test could be terminated if severe fatigue and extreme shortness of breath were experienced during the test.
  The results of the test were recorded.
Exercise Capacity | This test was carried out at baseline.
  The exercise capacity of the individuals was evaluated with the 6-Minute Walk Test (6 MWT), a submaximal test with high validity and reliability (ICC=0.94). 6MWT, made according to the American Thoracic Society guidlines.The distance covered in a 6-minute walk was calculated from the number of laps and meters. Values were recorded as a percentage of expected values for age and sex.
Exercise Capacity | This test was carried out at the 24th hours after DOMS.
  The exercise capacity of the individuals was evaluated with the 6-Minute Walk Test (6 MWT), a submaximal test with high validity and reliability (ICC=0.94). 6MWT, made according to the American Thoracic Society guidlines.The distance covered in a 6-minute walk was calculated from the number of laps and meters. Values were recorded as a percentage of expected values for age and sex.
Exercise Capacity | This test was carried out at 48th hours after DOMS.
  The exercise capacity of the individuals was evaluated with the 6-Minute Walk Test (6 MWT), a submaximal test with high validity and reliability (ICC=0.94). 6MWT, made according to the American Thoracic Society guidlines.The distance covered in a 6-minute walk was calculated from the number of laps and meters. Values were recorded as a percentage of expected values for age and sex.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Ozden, Principal Investigator — Cyprus International University, School of Physical Education and Sports; Ozge Ozalp, Study Director — Cyprus International University, Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation; Rabia Tugba Kilic, Study Director — Ankara Yildirim Beyazit University,Faculty of Health Sciences, Physiotherapy and Rehabilitation Department; Hayri Baran Yosmaoglu, Study Chair — Baskent University, Physiotherapy and Rehabilitation Department
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Yildirim Beyazit University,Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Ankara
  - Faculty of Health Sciences, Departmant of Physiotherapy and Rehabilitation, Baskent University, Ankara

REFERENCES:
- [Background] Benditt JO. Respiratory Care of Patients With Neuromuscular Disease. Respir Care. 2019 Jun;64(6):679-688. doi: 10.4187/respcare.06827. PMID 31110036
- [Background] Lieber RL, Friden J. Morphologic and mechanical basis of delayed-onset muscle soreness. J Am Acad Orthop Surg. 2002 Jan-Feb;10(1):67-73. PMID 11809052
- [Background] Imtiyaz S, Veqar Z, Shareef MY. To Compare the Effect of Vibration Therapy and Massage in Prevention of Delayed Onset Muscle Soreness (DOMS). J Clin Diagn Res. 2014 Jan;8(1):133-6. doi: 10.7860/JCDR/2014/7294.3971. Epub 2014 Jan 12. PMID 24596744
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692
- [Background] Jamurtas AZ, Theocharis V, Tofas T, Tsiokanos A, Yfanti C, Paschalis V, Koutedakis Y, Nosaka K. Comparison between leg and arm eccentric exercises of the same relative intensity on indices of muscle damage. Eur J Appl Physiol. 2005 Oct;95(2-3):179-85. doi: 10.1007/s00421-005-1345-0. Epub 2005 Jul 9. PMID 16007451
- [Background] Hotta N, Yamamoto K, Katayama K, Ishida K. The respiratory response to passive and active arm movements is enhanced in delayed onset muscle soreness. Eur J Appl Physiol. 2009 Feb;105(3):483-91. doi: 10.1007/s00421-008-0926-0. Epub 2008 Nov 15. PMID 19015869
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056